CLINICAL TRIAL: NCT03345303
Title: Bortezomib in Treating Patients With Intrahepatic Cholangiocellular Carcinoma Featuring PTEN Deficiency
Brief Title: Bortezomib in Intrahepatic Cholangiocellular Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhengang Yuan (Other)
Responsible Party: Sponsor-Investigator, Zhengang Yuan, Director of Oncology Department, Eastern Hepatobiliary Surgery Hospital
Organization: Eastern Hepatobiliary Surgery Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EHBH-201708
Record Dates: First submitted 2017-11-06; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Bortezomib
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Bortezomib

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bortezomib treatment (Experimental): 'Bortezomib Injectable Solution
  Interventions: Drug: Bortezomib
- supportive care (No Intervention): supportive care

INTERVENTIONS:
Drug: Bortezomib — Bortezomib Injectable Solution
  Other Names: velcade
  Arms: Bortezomib treatment

SUMMARY:
This study evaluates the efficacy and safety of second-line treatment of bortezomib in advanced intrahepatic cholangiocarcinoma patients.Half of participants will receive bortezomib while the other half will receive best supporting care.

DETAILED DESCRIPTION:
There's no standard second-line treatment for advanced intrahepatic cholangiocarcinoma patients.

Previous study indicated high mutation/deletion rate of PTEN gene in intrahepatic cholangiocarcinoma and poor prognosis of those patients with PTEN mutation/deletion. The investigators also found that the activity of proteasomes elevated in cholangiocarcinoma cells with PTEN mutation/deletion.

So the investigators suppose proteasomes inhibitor could improve prognosis of intrahepatic cholangiocarcinoma patients with PTEN mutation/deletion

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologic or cytologic diagnosis of intrahepatic cholangiocarcinoma with stage IV;
2. Have progressed after at least 2 cycles of systematic chemotherapy therapy（gemcitabine+cisplatin/gemcitabine+oxaliplatin）;
3. The previous treatment and the present trial registration must be at least 2 weeks apart, and they must have recovered from any toxicity of a previous treatment;
4. Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1;
5. Eastern Cooperative Oncology Group performance score (ECOG): 0-2; Life expectancy of at least 12 weeks;
6. Normal liver,kidney and bone marrow function；
7. Subjects who understand and voluntarily signed a written informed consent form.

Exclusion Criteria:

1. History of other malignancy within 3 years. Patients with central nervous system metastases or brain metastasis
2. There is any contraindication to use Bortezomib
3. Patients with contraindications (active bleeding, ulcers, intestinal perforation, intestinal obstruction, within 30 days after major surgery, uncontrolled high blood pressure medication, III-IV level cardiac insufficiency, severe liver and kidney dysfunction).
4. A previous history of Interstitial pulmonary disease, drug-induced interstitial disease, radiation pneumonitis requiring hormonal therapy or active interstitial lung disease with any clinical evidence.
5. Pregnant or lactating women.
6. History of radiation within 4 weeks prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | at least 2 months
  Objective response rate include response from stable disease to complete response based on RECIST 1.1

SECONDARY OUTCOMES:
changes of platelet count | 7 days
  changes of platelet count after injection of Bortezomib
occurrence of peripheral neuritis | 7 days
  occurrence of any feeling of numbness of limbs

CONTACTS AND LOCATIONS:
Locations (1):
- Easter hepatobiliary surgery hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zeng TM, Jiang TY, Yang G, Cheng Z, Lou C, Wei W, Tao CJ, Hu S, Wang H, Cui XW, Tan YX, Dong LW, Wang HY, Yuan ZG. Bortezomib in previously treated phosphatase and tension homology-deficient patients with advanced intrahepatic cholangiocarcinoma: An open-label, prospective and single-centre phase II trial. Clin Transl Med. 2024 May;14(5):e1675. doi: 10.1002/ctm2.1675. PMID 38689424